CLINICAL TRIAL: NCT01271166
Title: Glivec® Plus m-FOLFOX Avastin® in Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BAU14
Record Dates: First submitted 2011-01-04; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Advanced Colorectal Cancer
Keywords: Colorectal,; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Imatinib Mesylate; Fluorouracil; Oxaliplatin; Leucovorin; Bevacizumab

ARMS (1):
- Glivec®, modified FOLFOX, Avastin® (Experimental)
  Interventions: Drug: Imatinib, Fluorouracil, Oxaliplatin, Leucovorin and Bevacizumab

INTERVENTIONS:
Drug: Imatinib, Fluorouracil, Oxaliplatin, Leucovorin and Bevacizumab

SUMMARY:
This is a Phase I, dose finding, multicentre study evaluating the maximal tolerated dose of Glivec® in combination with mFOLFOX-Avastin®. Patients will be enrolled into each dose level in 3 patient cohorts. Additional cohorts will be enrolled, or dose levels opened, subject to the toxicities observed. Once the MTD has been determined the dose level below will be re-opened and extra patients, to a total of 15, will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally advanced, recurrent or metastatic colorectal cancer
* ECOG 0 or 1
* Measurable disease

Exclusion Criteria:

* Prior first line therapy for advanced disease
* Significant bulk of metastatic disease or rapid progression
* If prior adjuvant therapy, relapse within 6 months of a 5-FU based regimen or 12 months of an oxaliplatin based regimen

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Tumour response as assessed by CT scan and RESIST | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novarts Investigative Site, Melbourne, Australia